CLINICAL TRIAL: NCT07081685
Title: Efficacy of Non-Invasive Neuromodulation on Pain in Migraine
Acronym: ENDIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC I 2023 MOISSET; 2024-A01985-42 (Other: ANSM)
Record Dates: First submitted 2025-05-27; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-05

CONDITIONS: rTMS Stimulation; Migraine
Keywords: rTMS neurostimulation
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS stimulation (Experimental)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- sham rTMS stimulation (Sham Comparator)
  Interventions: Device: sham repetitive Magnetic Transcranial Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — robot-guided high-frequency rTMS treatment (10hz - 5 sessions) of the primary motor cortex
  Arms: rTMS stimulation
Device: sham repetitive Magnetic Transcranial Stimulation (rTMS) — sham robot-guided high-frequency rTMS treatment (10hz - 5 sessions) of the primary motor cortex
  Arms: sham rTMS stimulation

SUMMARY:
This is a prospective clinical study evaluating the analgesic efficacy of a non-medicated treatment: repeated transcranial magnetic stimulation (rTMS) of the primary motor cortex in chronic migraine (> 7 headache days per month and failure of at least 3 drug treatments).

To this end, the study involves a double-blind, randomized, comparative experimental protocol against a sham control condition via 2 parallel groups comprising 60 patients each (N= 120 in total). Randomized block design with stratification by center and type of migraine (episodic or chronic).

5 rTMS sessions will be performed, with one stimulation session every 2 weeks. One group will receive active stimulation at each session (high-frequency stimulation of the left primary motor cortex, 2000 pulses per session, 80% of resting motor threshold) and the other group placebo stimulation (sham).

Depending on the randomization group, rTMS sessions will be carried out by trained experimenters in the investigating center where the patient has been included. The study is multicentric, with five centers, four of which are in the Auvergne-Rhône-Alpes region. Data will be centralized at the Clermont-Ferrand University Hospital, and statistical analysis will be carried out by the Clermont-Ferrand University Hospital's Clinical Research and Innovation Department. Principal difference analysis (active vs sham) performed in ITT; missing data processed by multiple imputation.

ELIGIBILITY:
Inclusion criteria :

* Age greater than or equal to 18 years ;
* Frequent episodic or chronic migraine: migraine more than 8 days per month for more than 3 months;
* Maximum 26 headache days / 28 ;
* Failure (ineffectiveness, intolerance or contraindication) to at least 3 background drug treatments;
* Analgesic treatment stable for at least one month and will not need to be modified for the duration of the study;
* Patient can be followed throughout the study;
* Information letter read and understood;
* Signed informed consent;
* Affiliation with a social security scheme.

Exclusion Criteria:

* Contraindication to rTMS (patient with conductive/sensitive material to magnetic fields implanted in the skull or less than 30 cm from the coil, implanted material controlled by physiological signals, history of epilepsy or unexplained seizures, drug treatment lowering the epileptic threshold, brain lesions in relation to the stimulation zone [of vascular, traumatic, tumoral, infectious or metabolic origin], sleep deprivation, alcoholism, treatment with electroconvulsive therapy in the previous month, uncontrolled intracranial hypertension,
* Contraindication to MRI (ferromagnetic material not compatible with MRI including: intracerebral metal clip, pacemaker, insulin pump, intrathecal pump, metal prosthesis; severe claustrophobia)§ drug or psychoactive substance abuse
* Presence of other pain more severe than that justifying inclusion
* Patients under guardianship or deprived of liberty.
* Pregnant or breast-feeding women
* Patients participating in another research protocol involving a drug in the 30 days prior to inclusion.
* Subject having already benefited from rTMS sessions in the past (to maintain the blind)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Variation of headaches days number per month | difference between the 4 weeks prior to initiation of treatment and the last 4 weeks post-treatment

SECONDARY OUTCOMES:
variation in the number of headache (days per month) of at least 50% | between the 4 weeks prior to initiation of treatment and the last 4 weeks post-treatment
variation in the number of headache (days per month) of at least 30%. | between the 4 weeks prior to initiation of treatment and the last 4 weeks post-treatment
Patient Global Impression of Change (PGIC) | at week 12
  The score varies from 1 to 7 . A score of 1 means a better outcome and a score of 7 means a worse outcome

OTHER OUTCOMES:
Bang blinding index | week 0, week 2, week 4, week 6, week 8, week 12
  The patient will be asked what he thinks he received after the treatment, rTMS neuromodulation or sham neuromodulation
Variation of blood cytokine levels | Before (Week 0) and after treatment (Weeks 8 and 12)
  Following cytokines levels will be assessed : IL-6, IL-10, IL-17, IL-18, IL-1α, IL-1β, IL-21, IL-22, IL-23, IL-33, IL-35, CCL-20, IL-36β, IL-37, IL-38, IL-1Ra, TNFa, TGFβ, IL-2, INF-γ
Variation of headaches days number per month | Every each 4-week period post-treatment, compared to 4 weeks before treatment initiation
Migraine Hypersensitivity Assessment Questionnaire (MHQ-8 scale, ex-MIGAL) score | Pre-treatment period (inclusion visit at W0 - 4) and at week 12
  This scale assesses the frequency and intensity of disturbances related to noise, light, skin stimulation, and odors during migraines
Improvement in Quality of life by migraine rescue medication intakes | Week0 - 4 to week0 -1 period compared to Week 9 - week 12 period
  Improvement in quality of life will be assessed by use of migraine rescue medication before and after neurostimulation
Improvement in Quality of life by European Quality of Life 5 dimensions (EQ- 5D) scale score | At week 0, week 8 and week 12
  Improvement in quality of life will be assessed by the change of EQ-5D score
Improvement in Quality of life by relief subjective rate | At Week 2, week 4, week 6, week 8 and week 12
  A relief subjective rate since last neurostimulation will be asked to patient before each new neurostimulation session . A rate of 0% means "no relief" and 100% means a complete relief .
Improvement in Quality of life by anxiety and depression scores | At screening visit (Week 0 - 4) and week 12
  Anxiety and depression will be assessed by Hospital Anxiety and Depression Scale (HADS)
Improvement in Quality of life by resilience score | At screening visit (Week 0-4) and week 12
  Resilience score will be assessed by Connor-Davidson Resilience Scale (CD-RISC) in 25 items. The score ranges from 0 to 100 and a higher score means a higher resilience
Improvement in Quality of life by catastrophizing score | At screening visit (Week 0-4) and week 12
  Catastrophism will be assessed by Pain Catastrophizing Scale (PCS) . Score ranges from 0 to 52. A higher score indicates a higher level of catastrophizing of pain.
Improvement in Quality of life by intensity and emotional experience of pain | At screening visit (week 0- 4) and week 12
  A visual analogue scale (VAS) ranging from 0 to 100 for pain intensity and affective experience will be used.
Brain activity (resting-state fMRI) | At screening visit (week 0- 4) and week 12
  MRI recording is routinely carried out before any rTMS session. This involves acquiring a 3D image of the participants' brains, which is necessary for targeting cortical area stimulated by rTMS using a neuronavigation system. Functional imaging (fMRI) in a resting state (i.e., without a 'resting-state' task) will allow to measure the basal state of activity and connectivity in the participants' brains.
Cortical excitability | At week 0 and week 12
  measured during rTMS motor threshold with paired pulse stimulation measurements
Evaluation of side effects | up to 4 weeks post-treatment (at week 12)
Changes in prognostic markers of response | At week 0, week 8 and week 12
  Following blood parameters will be assessed : Blood count, CRP, Venous glycemia, Insulin, prolactin, estradiol, FSH, LH, progesterone, testosterone, β-hCG, CGRP, VIP, PACAP-38, IL-6, IL-10, IL-17, IL-18, IL-1α, IL-1β, IL-21, IL-22, IL-23, IL-33, IL-35, CCL-20, IL-36β, IL-37, IL-38, IL-1Ra, TNFa, TGFβ, IL-2, INF-γ, T lymphocyte immunophenotyping (CD3, CD4, CD25, FoxP3, CTLA-4, ICOS, TNFR2, CD45, CD45RA, CD8, CD14, 4-1-BB, NKp46, CD19, CD197, CD39, CD73, GITR, TCRaβ, CD127, CD56, CD62L)
Patient Global Impression of Change (PGIC) | week 2, week 4, week 6, week 8
  The score ranges from 1 to 7. A score of 1 means a better outcome and a score of 7 means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France, France

IPD SHARING:
Plan to Share IPD: No